CLINICAL TRIAL: NCT01128699
Title: Ahmed Valve Glaucoma Implant With Adjunctive Subconjunctival Bevacizumab in Refractory Glaucoma: a Randomized Controlled Clinical Trial
Brief Title: Ahmed Valve Glaucoma Implant With Adjunctive Subconjunctival Bevacizumab in Refractory Glaucoma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Vanak Eye Surgery Center (Other)
Responsible Party: Nader Nassiri, Associate Professor, Department of Ophthalmology, Imam Hossein Medical Center, Shaheed Beheshti University of Medical Sciences, Tehran, Iran
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VESC# 2010-142
Record Dates: First submitted 2010-05-21; First posted 2010-05-24 (Estimated); Last update posted 2010-05-24 (Estimated); Status verified 2010-05

CONDITIONS: Refractory Glaucoma
Keywords: Ahmed valve; Neovascular Glaucoma; Uveitic glaucoma; Failed glaucoma; VEGF-A; Intraocular pressure; Subconjunctival Avastin
MeSH Terms: conditions — Glaucoma; Glaucoma, Neovascular

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ISA+AVI (Experimental): injection of intraoperative subconjunctival Avastin as an adjunct to Ahmed valve implant
  Interventions: Drug: Subconjunctival Avastin
- AVI (Active Comparator): Ahmed valve implant
  Interventions: Device: Ahmed Valve implant

INTERVENTIONS:
Drug: Subconjunctival Avastin — Intraoperative Subconjunctival Avastin 1.25mg; single dose as an adjunct to 184 mm2 surface area Ahmed Glaucoma Valve (AGV Model FP7; New World Medical Inc., Rancho Cucamonga, California, USA)
  Arms: ISA+AVI
Device: Ahmed Valve implant — 184 mm2 surface area Ahmed Glaucoma Valve (AGV Model FP7; New World Medical Inc., Rancho Cucamonga, California, USA)
  Arms: AVI

SUMMARY:
The investigators aim to demonstrate the efficacy and safety of subconjunctival injection of Avastin as an adjunctive therapy for Ahmed valve glaucoma implant in patients with refractory glaucoma.

DETAILED DESCRIPTION:
Several studies have revealed evidences on the substantial role of Vascular endothelial growth factor-A (VEGF-A) in enhancing neovascularization processes. Some studies have shown the efficacy of intravitreal Avastin in reducing level of VEGF-A to improve NVG. On the other hand, recent pathological studies demonstrated that neutralization of VEGF reduced vascularity and decreased scar formation during wound healing, showing that VEGF strongly influence scar tissue formation. This may reduce the formation of encapsulated cyst after glaucoma surgeries and thus might improve the surgical success rate. The effect of subconjunctival bevacizumab as an adjunctive therapy in filtering glaucoma surgeries has been recently illustrated.

We aim to demonstrate the efficacy and safety of subconjunctival injection of Avastin as an adjunctive therapy for Ahmed valve glaucoma implant in patients with refractory glaucoma.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of refractory glaucoma defined as uncontrolled IOP (> 21 mm Hg) despite maximal antiglaucoma medication, previously failed surgical treatment, or a combination thereof

Exclusion Criteria:

* No light perception
* elevated IOP associated with silicone oil
* previous glaucoma drainage device implantation in the same eye
* previous cyclodestructive treatment
* increased risk of endophthalmitis (e.g., active adnexal and ocular surface infection, immunosuppression, or immunodeficiency, including the use of systemic steroids)
* posterior segment disorders, or pre-existing ocular comorbidities (e.g., pterygium, phacodonesis, corneal opacity, or corneal endothelial dystrophies).

Only 1 eye per patient was included in this trial.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2010-05; Primary Completion 2011-05 (Estimated); Study Completion 2011-07 (Estimated)

PRIMARY OUTCOMES:
Change in intraocular pressure (IOP) | 12 months
  To demonstrate the efficacy and safety of subconjuctival injection of Avastin as an adjunctive therapy for Ahmed valve glaucoma implant in patients with refractory glaucoma.

SECONDARY OUTCOMES:
Surgical failure | 12 months
Change in intraocular pressure | day 1, week 1, and months 1, 3, 6, 9

CONTACTS AND LOCATIONS:
Locations (1):
- Vanak Eye Surgery Center, Tehran, Iran